CLINICAL TRIAL: NCT03270930
Title: A Prospective Study of Evaluation of Operative Duration as a Predictor of Mortality in Pediatric Emergency Surgery: Concept of 100 Minutes Laparotomy in Resource-limited Setting
Brief Title: Operative Duration as a Predictor of Mortality in Pediatric Emergency Surgery
Status: Completed | Type: Observational
Sponsor: Jawaharlal Nehru Medical College (Other)
Responsible Party: Principal Investigator, Kaushal Deep Singh, Principal Investigator, Jawaharlal Nehru Medical College
Other Study IDs: JNMCH
Record Dates: First submitted 2017-08-23; First posted 2017-09-01 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Mortality; Pediatric; Laparotomy; Emergencies
Keywords: Operative duration; Pediatric surgery; Emergency laparotomy; Mortality rate; Survival; Kaplan-Meier analysis; ROC curve analysis; Senior resident
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survived: Pediatric patients in the age group of 5 to 10 years presenting with acute abdomen and undergoing emergency laparotomy who survived during their index 30-day hospital stay
  Interventions: Procedure: Emergency laparotomy
- Expired: Pediatric patients in the age group of 5 to 10 years presenting with acute abdomen and undergoing emergency laparotomy who expired during their index 30-day hospital stay
  Interventions: Procedure: Emergency laparotomy

INTERVENTIONS:
Procedure: Emergency laparotomy — All patients in study underwent emergency laparotomy within 24 hours of presentation after adequate resuscitation of minimum 1 hour.

SUMMARY:
Introduction Operative duration is an important but under-studied predictor of mortality in emergency laparotomies.

Aims & Objectives The objective of this study was to quantify the effect of duration of emergency laparotomy in children on mortality and to identify a rough cut-off duration of laparotomy to serve as a guide to plan the laparotomy to optimize pediatric surgical patient outcome.

DETAILED DESCRIPTION:
Operative duration has been found to affect post-operative mortality rates. Operative duration has been studied in various studies as a risk factor for predicting morbidity and several other post-operative complications like pneumonia. However, the direct effect of operative duration on mortality has been studied sparingly and that too mainly in elective setting and other authors. Thus, operative duration is an under-studied risk factor in predicting mortality in emergency laparotomies. No study was found during literature review which predicted mortality as a function of operative duration in emergency laparotomies. Most studies focused on pre-operative factors and post-operative management for predicting laparotomy outcomes like the use of POSSUM (Physiological and Operative Severity Score for the enumeration of Mortality and morbidity) score. Thus, no clear-cut recommendation exists regarding the optimal time duration for an emergency laparotomy in pediatric population beyond which a laparotomy must not proceed as it would significantly increase the mortality rate.

The primary objectives of the study were to quantify the effect of duration of emergency laparotomy in children on mortality and to identify a rough cut-off duration of laparotomy to serve as a guide so that such a laparotomy can be planned to optimize pediatric surgical patient out come in terms of decreased mortality. The secondary objectives included identifying factors that increase the time of emergency laparotomy and identifying measures that could be applied to reduce the time of laparotomy significantly and improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients in the age group of 5 to 10 years presenting with acute abdomen diagnosed clinically and radiologically to be having a diagnosis of secondary peritonitis and obstruction; who were adequately resuscitated (with a minimum resuscitation period of at least 1 hour) pre-operatively and underwent definitive surgery by a single surgeon (pediatric surgery senior resident) in the emergency were included in the study. Also, only those patients who had a PRISM-III (Pediatric Risk of Mortality III) score (Figure 1) of ≤ 8 at presentation were included to avoid the confounding effect of pre-operative variables that might affect mortality. All patients were adequately resuscitated in terms of temperature, central nervous system (Glasgow Coma Scale, pupillary reflexes), cardiovascular system (systolic blood pressure, heart rate) and respiratory system (oxygen saturation > 95%, pCO2 , pH, PaO2) parameters so that the patients were brought within 0 score range of PRISM-III score at the end of resuscitation and before shifting to the operation theatre. Furthermore for inclusion only those pediatric patients were considered who presented within 72 hours of initial onset of symptoms, operated within 24 hours of initial presentation and who died in index hospital admission within 30 days.

Exclusion Criteria:

* Patients who underwent damage control surgery, whose PRISM - III score was >9 at any point of time before undergoing laparotomy or inability to achieve adequate resuscitation (PRISM-III score >0 before shifting to operation theatre) and/or requirement of resuscitation beyond 4 hours of presentation were excluded from the study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients presenting to our emergency department in the age group of 5 to 10 years presenting with acute abdomen diagnosed clinically and radiologically to be having a diagnosis of secondary peritonitis and obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Effect of duration of laparotomy on pediatric post-operative mortality | 24 months
  This study primarily quantified the effect of duration of emergency laparotomy in children on mortality and also identified a rough cut-off duration of laparotomy as 100 minutes that such a laparotomy can be planned to optimize pediatric surgical patient out come in terms of decreased mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal D Singh, MS Surgery, Principal Investigator — Jawaharlal Nehru Medical College, Aligarh

IPD SHARING:
Plan to Share IPD: Yes
All the statistics of the patients like age, sex, operative duration, PRISM-III scores, duration of transfer to operation theatre and the final outcome will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available in the next 6 months and will be available for unlimited period of time
Access Criteria: Anyone can access the data here
URL: https://www.researchgate.net/project/Effect-of-Paediatric-Laparotomy-Operative-Duration-on-Mortality-in-Emergency-Surgeries

DOCUMENTS (3):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03270930/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03270930/SAP_001.pdf
  • Informed Consent Form (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03270930/ICF_002.pdf